CLINICAL TRIAL: NCT03747666
Title: Evaluating Masticatory Biting Force After Using Single Locking Miniplate Versus Two Non-locking Miniplates in the Management of Parasymphyseal Fracture in Patients With Two-line Mandibular Fractures
Brief Title: Single Locking Miniplate and Two Non-locking Miniplates in the Management of Parasymphyseal Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Abdelkader Hussein, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30101980
Record Dates: First submitted 2018-11-12; First posted 2018-11-20 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Mandible Fracture
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Locking miniplate (Experimental): The fractured segments in the parasymphyseal region will be fixed using 2.0 single locking miniplates and the fractured segments of the angle will be fixed conventionally using 2.0 single non-locking miniplate placed on the external oblique ridge.
  Interventions: Procedure: 2.0 single locking miniplates
- Non-locking miniplates (Experimental): The fractured segments in the parasymphyseal region will be fixed using 2.0 two non-locking miniplates and the fractured segments of the angle will be fixed conventionally using 2.0 single non-locking miniplate placed on the external oblique ridge.
  Interventions: Procedure: 2.0 single locking miniplates

INTERVENTIONS:
Procedure: 2.0 single locking miniplates — The fractured segments in the parasymphyseal region will be fixed using 2.0 single locking miniplates placed on the inferior border of the mandible.

SUMMARY:
Evaluating the biting force after management of parasymphyseal fracture in patients with two-line mandibular fractures.

DETAILED DESCRIPTION:
Evaluating the biting force after using 2.0 mm single locking miniplate versus 2.0 mm two conventional non-locking miniplates in the management of parasymphyseal fracture in patients with two-line mandibular fractures.

ELIGIBILITY:
Inclusion Criteria:

* Contra-lateral unfavorable non-comminuted simple or compound mandibular fracture in the parasymphyseal and angle regions.
* Fractures amenable to treatment using intra oral approach.

Exclusion Criteria:

* Medically compromised patients who are unfit for the procedure under general anesthesia.
* Patients with comminuted fractures.
* Patients with history of occlusion disturbances or skeletal malocclusion.
* Patients with insufficient dentition to reproduce occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Biting force | 6 months
  Biting force will be measured using occlusal biting force meter (Higher biting force record is better)

SECONDARY OUTCOMES:
Stability of fractured segments | 6 weeks
  Bi-manual manipulation (Binary Yes/No)
Pain intensity | 10 days
  Visual analog scale (0-10) 0=No pain & 10=Severe pain
Occlusion | 6 months
  Clinical examination (Intact/Deranged)
Infection | 6 months
  Clinical examination (Present/Absent)
Hardware failure | 6 months
  Clinical examination (Present/Absent)
Paraesthesia | 6 months
  Observation/Contact detection/Pin-brick nociception (0-10) 0=No sensation & 10= Normal sensation
Wound dehiscence | 6 months
  Clinical examination (Present/Absent)